CLINICAL TRIAL: NCT05763043
Title: Monoferric for Prenatal Iron Deficiency
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ashley Benson, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB 25397
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obstetric Labor Complications
MeSH Terms: conditions — Obstetric Labor Complications | interventions — ferric derisomaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferric derisomaltose (Experimental)
  Interventions: Drug: Ferric derisomaltose

INTERVENTIONS:
Drug: Ferric derisomaltose — Participants between the gestational ages of 14 to 42 weeks with iron deficiency will receive IV Ferric derisomaltose at a routine prenatal visit.
  Other Names: Monoferric

SUMMARY:
A prospective observational study of pregnant women with iron deficiency anemia and oral iron intolerance or advanced gestational age.

DETAILED DESCRIPTION:
Intravenous therapy (IV) Monoferric (ferric derisomaltose), is a single-dose, rapid infusion formulation that has the potential to reduce both time and cost barriers, though its efficacy and safety in pregnant women has not been well studied. Thus, we propose to study the safety and efficacy of single dose, monoferric 1,000 mg IV in a cohort of pregnant participants with iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years of age or older between 14 to 42 weeks gestation who are deemed appropriate for IV iron by their treating provider as part of their standard of care treatment.
* Iron deficiency anemia, defined as second or third trimester (14 weeks or more) hemoglobin less than or equal to 10.5 g/dL or less than or equal to11 g/dL, respectively, and ferritin less than 50 μg/L
* Experience intolerance to oral iron or are greater than 28 weeks gestation
* Willing to participate in the study

Exclusion Criteria:

* Known infectious, inflammatory, or malignant conditions that may confound iron repletion and outcome analysis
* Prior IV iron intolerance or hypersensitivity reaction

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who experienced a resolution of iron deficiency anemia | From enrollment to 6 weeks post partum
  The proportion of participants who experienced a resolution of iron deficiency anemia, defined as a 1 g/dL increase in Hgb at a follow up assessment at 6 weeks postpartum following IV Monoferric administration

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science Univerity, Portland, Oregon, United States